CLINICAL TRIAL: NCT02308215
Title: Retinal Therapy Guided by 3D OCT Image Analysis
Status: Completed | Type: Observational
Sponsor: Michael Abramoff (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor-Investigator, Michael Abramoff, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201003712; 1R01EY019112-01A2 (NIH)
Record Dates: First submitted 2014-11-13; First posted 2014-12-04 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Age-Related Macular Degeneration; Choroidal Neovascularization
Keywords: Retina; AMD; OCT
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose is to find a better way to predict the timing of treatments given to patients with Wet Age-related macular degeneration using image analysis.

DETAILED DESCRIPTION:
The study focuses on making better use of advanced three-dimensional imaging and analysis to allow physicians to know when a treatment is being effective and thus not overuse it. The study will examine how 3-D optical coherence tomography and related image analysis can be used to assess changes in the macula and retina of patients' eyes. These changes can reveal how well a person is responding to anti-VEGF treatment and thus help doctors provide proper treatment timing and care.

ELIGIBILITY:
Inclusion Criteria:

* fundoscopically confirmed AMD and patient eligible for treatment with anti-VEGF

Exclusion Criteria:

* Patients with a CNV due to other causes (OHS, trauma)
* eyes that have been previously treated for CNV

Ages: 45 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed research will be carried out in patients diagnosed with Choroidal Neovascularization associated with AMD selected from retina care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2010-07; Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Measure central retinal layer thickness in µms. | one year
Measure amount of fluid in the retina in µms. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Abramoff, MD, PhD, Principal Investigator — University of Iowa; Milan Sonka, MS, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals Dept of Ophthalmology, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No